CLINICAL TRIAL: NCT03353207
Title: Striatal Dopamine Transmission in Individuals With Isolated Rapid Eye Movement Sleep With Atonia: a Search for Precursor Biomarker for Neurodegeneration
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: HMRF04153036
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: REM Sleep Behavior Disorder; Neurodegenerative Diseases
Keywords: REM Sleep Without Atonia; Dopamine transmission; Neurodegeneration
MeSH Terms: conditions — REM Sleep Behavior Disorder; Neurodegenerative Diseases; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- health Control: 1. No family history of RBD;
  2. Age- and sex- matched with isolated RSWA subjects
  3. Absence of dream enactment behaviors;
  4. A score of RBDQ-HK less than 19;
  5. Absence of RSWA as measured by v-PSG;
  6. for those individuals with moderate obstructive sleep apnea (AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.
- Case with isolated RSWA: 1. First degree relatives of patients with iRBD;
  2. Age 45 years or above;
  3. Absence of dream enactment behaviors;
  4. A total score on REM Sleep Behavior Questionnaire (RBDQ-HK) less than 19, which is the cut-off suggestive of a diagnosis of RBD;
  5. Presence of RSWA as measured by v-PSG; RSWA is defined as the percentage of increased EMG activity (phasic or tonic) at least 10% during REM sleep for any channel.
  6. for those individuals with moderate to severe obstructive sleep apnea (apnea-hypopnea index, AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.
- Case without isolated RSWA: 1. First degree relatives of patients with iRBD;
  2. Age- and sex- matched with isolated RSWA subjects;
  3. Absence of dream enactment behaviors;
  4. A score of RBDQ-HK less than 19;
  5. Absence of RSWA as measured by v-PSG;
  6. for those individuals with moderate obstructive sleep apnea (AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.

SUMMARY:
Background:

Previous studies have confirmed that most patients with idiopathic REM sleep behaviour disorder (iRBD) eventually develop neurodegenerative diseases. In addition, REM sleep without atonia (RSWA), a hallmark of RBD feature, is a significant predictor of development of neurodegenerative diseases in patients with iRBD. Some preliminary studies have implied that isolated RSWA in the absence of RBD symptoms may also indicate neurodegeneration. However, this speculation needs to be confirmed by more refined study with sophisticated measures in both RSWA and markers of neurodegeneration

Objectives: 1) to determine the differences in striatal dopamine transmission and other markers of neurodegeneration among individuals with isolated RSWA and healthy controls; 2) to examine the correlation of severity of RSWA with striatal dopamine transmission.

Design: Case-control study

Setting: Community-based sample

Participants: 1) iRBD first degree relatives with isolated RSWA (n=18) 2) iRBD first degree relatives without isolated RSWA (n=18) 3) Community-based health controls without isolated RSWA (n=18)

Main outcome measures:

1. The dopamine transmission as measured by triple-tracer PET/ CT imaging protocol including 18F-DOPA, 11C-Raclopride and 18F-FDG images;
2. Brain glucose metabolism and neurocognitive measures;
3. Severity of EMG activity during REM sleep

DETAILED DESCRIPTION:
In the past two decades, a number of studies have confirmed that most patients with idiopathic RBD will eventually develop neurodegenerative diseases, especially α-synucleinopathies. Previous studies, including our preliminary data, suggested that RSWA is a marker of predicting the conversion of neurodegenerative diseases in idiopathic RBD. In other words, RSWA is an early marker of neurodegeneration in patients with idiopathic RBD. However, a number of individuals who are absent of any RBD symptoms (including patients with α-synucleinopathies, also have RSWA, which is described to have isolated RSWA. Only a few studies have attempted to understand the clinical importance and predictive prognosis of isolated RSWA. These preliminary studies suggest that isolated RSWA in healthy subjects may be a silent biomarker of neurodegeneration. However, these preliminary findings need to be replicated and confirmed by more refined study with dopamine neurotransmission neuroimaging.

This proposed study will enrich the limited scientific literature of the potential pathogenesis and progression of isolated RSWA. By using an ongoing family study, we have screened a number of individuals with isolated RSWA, who are the first degree relatives of patients with RBD and are presumed to have a higher risk of neurodegeneration. Based on the existing sample, the current study will provide the first neuroimaging data on isolated RSWA to test the hypothesis that isolated RSWA, even in the absence of RBD symptoms, is an early marker of neurodegeneration. Individuals with isolated RSWA are expected to show dopamine dysfunction when compared with individuals without RSWA. If we confirm this hypothesis, the findings in the current study will extend our understanding of the spectrum of RBD and RSWA. The potential implication of our findings is that asymptomatic RSWA, especially in the presence of family history, will harbour the neurodegenerative progression. The results will pave the way for future prospective follow up to determine the course of neurodegeneration. From an etiological understanding, it will help to expand the understanding of the evolution course of synucleinopathy neurodegeneration. From an interventional angle, this study will have significant implication for developing a longer prevention window for neuroprotective trial.

The inclusion criteria for the subjects:

iRBD first degree relatives with isolated RSWA

1. First degree relatives of patients with iRBD;
2. Age 45 years or above;
3. Absence of dream enactment behaviors;
4. A total score on REM Sleep Behavior Questionnaire (RBDQ-HK) less than 19, which is the cut-off suggestive of a diagnosis of RBD;
5. Presence of RSWA as measured by v-PSG; RSWA is defined as the percentage of increased EMG activity (phasic or tonic) at least 10% during REM sleep for any channel.
6. for those individuals with moderate to severe obstructive sleep apnea (apnea-hypopnea index, AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.

Community-based health controls without isolated RSWA:

1. No family history of RBD;
2. Age- and sex- matched with isolated RSWA subjects
3. Absence of dream enactment behaviors;
4. A score of RBDQ-HK less than 19;
5. Absence of RSWA as measured by v-PSG;
6. for those individuals with moderate obstructive sleep apnea (AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.

ELIGIBILITY:
Inclusion Criteria:

1. No family history of RBD;
2. Age- and sex- matched with isolated RSWA subjects
3. Absence of dream enactment behaviors;
4. A score of RBDQ-HK less than 19;
5. Absence of RSWA as measured by v-PSG;
6. for those individuals with moderate obstructive sleep apnea (AHI > 15/hour), effective CPAP treatment should be documented and a second night of V-PSG is required to determine RSWA.

Exclusion Criteria:

1. Presence of dream enactment behaviors by self-report or documented by v-PSG;
2. Presence of narcolepsy and other neurological diseases that may give rise to RBD and RWSA;
3. Presence of neurodegenerative diseases;
4. A total score of the MOCA ≤ 22 and the CDR ≥ 1.
5. On medication that potentially increases EMG activity and triggers the symptoms of RBD, such as antidepressants;
6. On medication that affects dopamine neural transmission;
7. Not capable of giving informed consent for participation of the study.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified and recruited from our previous cohort.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Dopamine neurotransmission | 24 months
  PET dopamine neurotransmission with a specific interest in striatal dopamine transmission

SECONDARY OUTCOMES:
REMREEA | 24 months
  Correlations of severity of REMREEA with dopamine transmission, brain glucose metabolism, and neurocognitive measures.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Shatin Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
In this stage, we didin't decide which information of IPD will share with other researchers